CLINICAL TRIAL: NCT01240447
Title: A Prospective, Randomised, Open Label Phase II Study of Active Specific Immunotherapy With Racotumomab Versus Support Treatment in Patients With Advanced Non-small Cell Lung Cancer
Brief Title: Immunotherapy With Racotumomab Versus Support Treatment in Advanced Non-small Cell Lung Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Laboratorio Elea Phoenix S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AR-RACO-02-08; ISRCTN47153584 (Registry Identifier: Intl Standard Randomised Controlled Trial Number Register)
Record Dates: First submitted 2010-09-23; First posted 2010-11-15 (Estimated); Last update posted 2014-07-10 (Estimated); Status verified 2014-07

CONDITIONS: Advanced Non-small Cell Lung Cancer
Keywords: NSCLC; lung cancer, small-cell; advanced lung cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — racotumomab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Best support treatment (Other)
  Interventions: Other: Best support treatment
- Racotumomab vaccine (Experimental)
  Interventions: Biological: racotumomab

INTERVENTIONS:
Biological: racotumomab — Patients will receive best support treatment and vaccination with racotumomab. The vaccination schedule is as follows: 5 doses (1mg/mL each), subcutaneously, every 2 weeks (induction period) followed by monthly vaccinations until any criteria for discontinuation are met. If disease progression occurs and a second line therapy is indicated, the patient will only be able to continue in the study if the drug indicated is docetaxel. Vaccination will not be interrupted during docetaxel administration unless criteria for vaccine discontinuation are met.
  Other Names: 1E10
  Arms: Racotumomab vaccine
Other: Best support treatment — Patients will receive best support treatment as indicated by the investigator. In case a second line therapy is indicated, docetaxel is the only drug allowed to continue in the study.
  Arms: Best support treatment

SUMMARY:
This study is designed to evaluate safety and immunogenicity of racotumomab in patients with advanced Non-small Cell Lung Cancer (NSCLC), in concomitance with chemotherapy (docetaxel) when a second-line therapy is indicated. The study will also compare survival and progression free survival on both study arms.

ELIGIBILITY:
Inclusion Criteria:

1. The patient (aged over 21 years, either sex) can comply with the protocol and scheduled appointments and sign voluntarily the informed consent form
2. Diagnosis of Non-small cell lung cancer (NSCLC) stages IIIA (surgically unresectable), IIIB or IV, according to the TNM classification (Tumor-Nodes-Metastases) version 6a, confirmed by cytology or histology, if possible available for determination of ganglioside expression
3. Patients may enter the study if they have accomplished an objective response (complete response or partial response) or disease stabilisation (by Response Evaluation Criteria In Solid Tumours [RECIST]) after completion of standard onco-specific treatment. In all cases, response should be documented.

   For stage IIIA and IIIB without pleural effusion ("dry IIIB") standard treatment is considered as follows: 2 - 4 cycles of platinum-based chemotherapy and/or radiotherapy with curative intent in accordance with National Comprehensive Cancer Network (NCCN) guidelines For stage IIIB with pleural effusion ("wet IIIB") and stage IV standard treatment is considered as follows: 4 - 6 cycles of chemotherapy based on platinum. In case of pleural or pericardial effusion requiring local treatment, it will be provided prior to study entry.
4. Patients with an interval greater than 30 and not more than 90 days between the completion of oncospecific treatment and study entry. Completion of treatment is defined as the last day of administration of chemotherapy or the last day of radiotherapy. Patients should have recovered from any related episode of acute toxicity of degree greater than 1 (except alopecia). Patients who have received a monoclonal antibody (eg bevacizumab) should also have discontinued its use for at least 30 days before inclusion.
5. The subject is male or female, aged greater than or equal to 21 years
6. Performance status (Eastern Cooperative Oncology Group [ECOG]) less than or equal to 1
7. Acceptable organ functionality as defined by the following parameters:

   * Electrocardiogram (ECG) without significant abnormalities, performed within 14 days prior to admission
   * Haemoglobin greater than or equal to 90 g/L
   * Total leukocyte count greater than or equal to 3.0 x 10^9/L
   * Absolute neutrophil count greater than or equal to 1.5 x 10^9/L
   * Total bilirubin less than or equal to 1.5 times upper limit of normal or twice the limit normal than in case liver metastases are present
   * Serum glutamic oxaloacetic transaminase (SGOT) and serum glutamic pyruvic transaminase (SGPT) less than or equal to 2.5 times upper limit of normal (less than or equal to five times the normal maximum in case liver metastases are present)
   * Creatinine less than or equal to 2 mg/dL
8. Life expectancy of at least four months

Exclusion Criteria:

1. Patient is pregnant or breastfeeding
2. Has received chemotherapy, radiotherapy, immunotherapy or surgery within 30 days prior to inclusion
3. Hypersensitivity to any component of the formulation
4. Patients of childbearing potential of either sex who are not using an adequate method of contraception during treatment to avoid pregnancy (own or of partner). For females: intrauterine devices, hormonal contraceptives, barrier methods or sterilisation. For males: vasectomy or condoms with spermicide.
5. Patients receiving or having received other investigational drugs 30 days prior to study entry
6. History of autoimmune diseases
7. Decompensated chronic diseases
8. Acute allergic disorders or history of severe allergic reactions
9. Known brain metastases uncontrolled with surgery and/or radiation therapy or under current corticosteroid therapy
10. History of inflammatory or demyelinating disease of the central or peripheral nervous system
11. Uncontrolled intercurrent illnesses, including active infection, symptomatic congestive heart failure, unstable angina or cardiac arrhythmia and psychiatric diseases implying patient incompetence
12. Other malignancies, with the exception of basal cell carcinoma, in situ cervical carcinoma, incidental prostate cancer (T1a, Gleason less than or equal to 6, prostate specific antigen [PSA] less than 0.5 ng/ml), tumour or any other tumour adequately treated and with a disease-free period greater than or equal to 5 years
13. Chronic treatment with systemic corticosteroids at doses greater than 0.5 mg/kg/day or a maximum of 40 mg/day of prednisone or equivalent
14. The subject has a history of drug abuse (illicit drugs) or alcohol abuse (defined as regular or periodic ingestion of more than four drinks a day) in the last 2 years
15. Positive serology for hepatitis B, C or known human immunodeficiency virus (HIV) infection
16. Uncontrolled hypercalcaemia greater than or equal to 2.9 mmol/L (or grade greater than 1 according to the Common Terminology Criteria for Adverse Events [CTCAE] version 3.0)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2009-09; Primary Completion 2012-08 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse events as a measure of safety and tolerability | Until death, on average during 17 months
  Safety will be evaluated at each study visit according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 3.0 and will include physical examination with vital signs, performance status as per the Eastern Cooperative Oncology Group scale(ECOG scale), laboratory tests and clinical history.
Evaluation of the reactivity if the antibodies against X63 tumor line | Baseline
Determination of T supressor cell (Treg cell) frequency by immunostaining and flow cytometry. | Baseline
Evaluation of the reactivity of the antibodies against the patients tumoral tissue (whenever samples are available) | Baseline
Determination of gamma interferon by ELISPOT (enzyme-linked immunosorbent spot) assay. | Baseline
Measurement of pro-inflammatory and anti-inflammatory cytokines | Baseline
Determination of T supressor cell (Treg cell) frequency by immunostaining and flow cytometry. | Month 2
Determination of T supressor cell (Treg cell) frequency by immunostaining and flow cytometry. | Month 4
Determination of T supressor cell (Treg cell) frequency by immunostaining and flow cytometry. | Month 8
Determination of T supressor cell (Treg cell) frequency by immunostaining and flow cytometry. | Month 12
Determination of IgM and IgG antibody titers against N-Glycolil-GM3 ganglioside | Baseline
Evaluation of the reactivity of the antibodies against the patients tumoral tissue (whenever samples are available) | Month 2
Measurement of pro-inflammatory and anti-inflammatory cytokines. | Baseline
Determination of IgM and IgG antibody titers against N-Glycolil-GM3 ganglioside | Month 2
Determination of IgM and IgG antibody titers against N-Glycolil-GM3 ganglioside | Month 8
Determination of IgM and IgG antibody titers against N-Glycolil-GM3 ganglioside | Month 4
Determination of IgM and IgG antibody titers against N-Glycolil-GM3 ganglioside | Month 12
Determination of IgM and IgG antibody titers against N-Glycolil-GM3 ganglioside | Every 4 months (after the first year, on average during 17 months)
Evaluation of the reactivity if the antibodies against X63 tumor line | Month 2
Evaluation of the reactivity if the antibodies against X63 tumor line | Month 12
Evaluation of the reactivity if the antibodies against X63 tumor line | Every 4 months (after the first year, on average during 17 months)
Evaluation of the reactivity if the antibodies against X63 tumor line | Month 4
Evaluation of the reactivity if the antibodies against X63 tumor line | Month 8
Evaluation of the reactivity of the antibodies against the patients tumoral tissue (whenever samples are available) | Month 4
Evaluation of the reactivity of the antibodies against the patients tumoral tissue (whenever samples are available) | Month 8
Evaluation of the reactivity of the antibodies against the patients tumoral tissue (whenever samples are available) | Month 12
Evaluation of the reactivity of the antibodies against the patients tumoral tissue (whenever samples are available) | Every 4 months (after the first year, on average during 17 months)
Determination of gamma interferon by ELISPOT (enzyme-linked immunosorbent spot) assay. | Month 2
Determination of gamma interferon by ELISPOT (enzyme-linked immunosorbent spot) assay. | Month 4
Determination of gamma interferon by ELISPOT (enzyme-linked immunosorbent spot) assay. | Month 8
Determination of gamma interferon by ELISPOT (enzyme-linked immunosorbent spot) assay. | Month 12
Determination of gamma interferon by ELISPOT (enzyme-linked immunosorbent spot) assay. | Every 4 months (after the first year, on average during 17 months)
Measurement of pro-inflammatory and anti-inflammatory cytokines | Month 2
Measurement of pro-inflammatory and anti-inflammatory cytokines | Month 4
Measurement of pro-inflammatory and anti-inflammatory cytokines | Month 8
Measurement of pro-inflammatory and anti-inflammatory cytokines | Month 12
Measurement of pro-inflammatory and anti-inflammatory cytokines | Every 4 months (after the first year, on average during 17 months)

SECONDARY OUTCOMES:
Survival | Until date of death or last censored observation
  On average, during 17 months
Progression free survival | Until first progression of disease
  Tumour evaluations will be performed every 2 months and evaluated as per Response Evaluation Criteria in Solid Tumors (RECIST).

CONTACTS AND LOCATIONS:
Overall Officials: Gabriela Cinat, MD, Principal Investigator — Instituto de Oncología "Angel H. Roffo"
Locations (1):
- Instituto de Oncología "Angel H. Roffo", Buenos Aires, Buenos Aires, Argentina